CLINICAL TRIAL: NCT00586612
Title: Immunogenicity & Safety Study in Preterm & Full-term Infants of GSK Biologicals' Hib-MenC Vaccine, Menitorix™ Co-administered With Infanrix™ Penta & Prevenar™ at 2, 4, 6 Months & as a Booster With Infanrix™ IPV & Prevenar™ at 16-18 Months
Brief Title: Primary & Booster Study to Evaluate the Immunogenicity and Safety of Menitorix Vaccine in Preterm Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110215; 110217 (Other: GSK)
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2010-01-22 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2016-10

CONDITIONS: Haemophilus Influenzae Type b; Neisseria Meningitidis
Keywords: Conjugate vaccine; Persistence; Hib vaccine; Combination vaccine; Meningococcal vaccine; Safety; Preterm/full-term infants; Immunogenicity
MeSH Terms: conditions — Haemophilus Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

ARMS (2):
- Preterm group (Experimental): Subjects born after a gestation period of less than or equal to 36 weeks and who received 3 doses (at 2, 4 and 6 months of age) of Menitorix™, Infanrix™ penta and Prevenar™ and a booster dose of Menitorix™, Infanrix™ IPV and Prevenar™ at 16-18 months of age.
  Interventions: Biological: Menitorix™; Biological: Infanrix™ penta; Biological: Prevenar™; Biological: Infanrix™ IPV
- Full-term group (Active Comparator): Subjects born after a gestation period of more than 36 weeks and who received 3 doses (at 2, 4 and 6 months of age) of Menitorix™, Infanrix™ penta and Prevenar™ and a booster dose of Menitorix™, Infanrix™ IPV and Prevenar™ at 16-18 months of age.
  Interventions: Biological: Menitorix™; Biological: Infanrix™ penta; Biological: Prevenar™; Biological: Infanrix™ IPV

INTERVENTIONS:
Biological: Menitorix™ — Intramuscular injection, 3 doses in the primary study and 1 dose in the Booster study.
Biological: Infanrix™ penta — Intramuscular injection, 3 doses in the primary study
Biological: Prevenar™ — Intramuscular injection, 3 doses in the primary study and 1 dose in the Booster study.
Biological: Infanrix™ IPV — Intramuscular injection, 1 dose in the Booster study.

SUMMARY:
The purpose of this Phase IIIb study is to evaluate the immunogenicity, reactogenicity & safety of GSK Biologicals' Hib-MenC vaccine (Menitorix™) when co-administered with GSK Biologicals' DTPa-HBV-IPV vaccine (Infanrix™ penta) & Wyeth's 7-valent pneumococcal conjugate vaccine (Prevenar™) in preterm infants as a 3-dose primary vaccination course during the first 6 months of life (at 2, 4, 6 months of age) and of a booster dose of Menitorix™ when co-administered with GSK Biologicals' DTPa-IPV vaccine (Infanrix IPV) and Wyeth's Prevenar in the second year of life (16-18 months of age). The control is a group of full-term infants receiving the same vaccines. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
This multicenter study is open & consists of a primary & a booster phase. The study has 2 treatment groups (Preterm & Full-term) that will receive the same vaccinations; the Full-term group will be the active control. Four blood samples will be collected from all subjects for immunogenicity analyses; 2 in the primary phase at prior to the first vaccination and one month after the third vaccination and 2 in the booster phase at prior to booster dose and one month after booster dose.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at study entry:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* A male or female between, and including, 8 and 12 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.

All preterm subjects must satisfy the following criteria at study entry:

* Born after a gestation period of less than or equal to 36 weeks (≤258 days).
* Medically stable, i.e. do not require significant medical support or ongoing management for debilitating disease and have demonstrated a clinical course of sustained recovery.

All full-term subjects must satisfy the following criteria at study entry:

* Born after a gestation period between and including 37 and 42 weeks (≥259 days and ≤294 days).
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration/ administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose of vaccine until the last study visit, except measles-mumps-rubella (MMR) and varicella vaccines which may be given according to local immunisation practices and except rotavirus oral vaccine which is allowed at anytime during the study after hospital discharge as per prescribing information.
* Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b, meningococcal serogroup C and or Streptococcus pneumoniae disease, with the exception of hepatitis B vaccine or BCG vaccine given in the first month of life according to the national recommendations (although BCG and hepatitis B vaccines should have been given outside a 30-day window from the first administration of study vaccines).
* History of diphtheria, tetanus, pertussis, polio, hepatitis B, H. influenzae type b, meningococcal disease and or S. pneumoniae disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins (with the exception of monoclonal antibodies against respiratory syncytial virus [RSV]) and/or any blood products within one month (30 days) preceding the first dose of study vaccines.
* Planned administration of immunoglobulins and/or any blood products during the active phase of the study.

Specific criteria for the booster part of the study (to be checked at Visit 5, study month 14):

* History of diphtheria, tetanus, pertussis, polio, hepatitis B, H. influenzae type b, meningococcal disease and or S. pneumoniae disease.
* Previous vaccination, except the study vaccines and hepatitis birth dose, against diphtheria, tetanus, pertussis, polio, hepatitis B, H. influenzae type b, meningococcal disease and or S. pneumoniae disease.
* Previous booster vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, H. influenzae type b, meningococcal disease and/or S. pneumoniae disease.

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 313 (Actual)
Dates: Start 2007-12-01; Primary Completion 2008-12-30 (Actual); Study Completion 2008-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Burgos
  - GSK Investigational Site, Getafe
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Móstoles/Madrid

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 110215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study are summarised with 110217 on the GSK Clinical Study Register.
- Available data/document: Informed Consent Form: 110215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 110215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110215 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Primary Phase
Arm/Group | Preterm Group | Full-term Group
Started | 163 | 150
Completed | 162 | 147
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Period: Booster Phase
Arm/Group | Preterm Group | Full-term Group
Started | 154 | 144
Completed | 151 | 143
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preterm Group | Full-term Group | Total
Number analyzed (Participants) | 163 | 150 | 313
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 8.9 (1.15) | 8.8 (0.79) | 8.9 (0.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 65 | 142
  Male | 86 | 85 | 171

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentration Greater Than or Equal to 0.15 Micrograms Per Milliliter (µg/mL)
Description: Anti-PRP antibody concentration greater than or equal to 0.15 µg/mL is indicative of protection.
Time Frame: One month after the third vaccination
Population: Analysis was performed on the Primary According-to-Protocol (ATP) cohort for immunogenicity, on subjects with available data.
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 140 | 142
subjects | 139 | 141

2. Primary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titer Greater Than or Equal to 1:8
Description: rSBA-MenC titer greater than or equal to 1:8 is indicative of protection.
Time Frame: One month after the third vaccination
Population: Analysis was performed on the Primary According-to-Protocol (ATP) cohort for analysis of immunogenicity, on subjects with available data.
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 143 | 140
subjects | 142 | 140

3. Secondary Outcome: Number of Subjects With Anti-Polyribosylribitol Phosphate (Anti-PRP) Antibody Concentration Greater Than or Equal to the Cut-off Values
Description: Anti-PRP antibody cut-off values assessed include 0.15 micrograms per milliliter (µg/mL) and 1 µg/mL.
Time Frame: Before vaccination (at Day 0)
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 140 | 138
subjects
  ≥ 0.15 µg/mL | 38 | 43
  ≥ 1.0 µg/mL | 5 | 9

4. Secondary Outcome: Number of Subject With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentration Greater Than or Equal to 1 Microgram Per Milliliter
Description: Anti-PRP antibody cut-off value assessed include 1 microgram per milliliter (µg/mL).
Time Frame: One month after the third vaccination
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 140 | 142
subjects | 133 | 134

5. Secondary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titer Greater Than or Equal to the Cut-off Values
Description: rSBA-MenC titer cut-off values assessed include 1:8, 1:32 and 1:128.
Time Frame: Before vaccination (at Day 0)
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 141 | 137
subjects
  ≥ 1:8 | 16 | 23
  ≥ 1:32 | 5 | 11
  ≥ 1:128 | 0 | 3

6. Secondary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titer Greater Than or Equal to the Cut-off Values
Description: rSBA-MenC titer cut-off values assessed include 1:32 and 1:128.
Time Frame: One month after the third vaccination
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 143 | 140
subjects
  ≥ 1:32 | 142 | 139
  ≥ 1:128 | 135 | 136

7. Secondary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC) Antibody Concentration Greater Than or Equal to (≥) the Cut-off Values
Description: Anti-PSC antibody cut-off values assessed include 0.3 micrograms per milliliter (µg/mL) and 2 µg/mL.
Time Frame: Before vaccination (at Day 0)
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 142 | 137
subjects
  ≥ 0.3 µg/mL | 23 | 36
  ≥ 2.0 µg/mL | 3 | 8

8. Secondary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC) Antibody Concentration Greater Than or Equal to (≥) the Cut-off Values
Description: Anti-PSC antibody cut-off values assessed include 0.3 micrograms per milliliter (µg/mL) and 2 µg/mL.
Time Frame: One month after the third dose
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 140 | 141
subjects
  ≥ 0.3 µg/mL | 140 | 141
  ≥ 2.0 µg/mL | 127 | 136

9. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration Greater Than or Equal to (≥) the Cut-off Values
Description: Anti-HBs antibody cut-off values assessed include 10 milli-international units per milliliter (mIU/mL) and 100 mIU/mL.
Time Frame: Before vaccination (at Day 0)
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 112 | 118
subjects
  ≥ 10 mIU/mL | 89 | 78
  ≥ 100 mIU/mL | 3 | 8

10. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration Greater Than or Equal to (≥) the Cut-off Values
Description: Anti-HBs antibody cut-off values assessed include 10 milli-international units per milliliter (mIU/mL) and 100 mIU/mL.
Time Frame: One month after the third dose
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 129 | 129
subjects
  ≥ 10 mIU/mL | 128 | 129
  ≥ 100 mIU/mL | 109 | 117

11. Secondary Outcome: Anti-polyribosylribitol Phosphate (Anti-PRP) and Anti-polysaccharide C (Anti-PSC) Concentration
Description: Anti-PRP and anti-PSC concentrations are given as geometric mean concentrations (GMCs) expressed micrograms per milliliter (µg/mL).
Time Frame: Before vaccination (at Day 0)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per milliliter (µg/mL)
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 142 | 138
micrograms per milliliter (µg/mL)
  Anti-PRP (n=140, 138) | 0.116 [0.101 to 0.133] | 0.140 [0.117 to 0.167]
  Anti-PSC (n=142, 137) | 0.19 [0.17 to 0.22] | 0.25 [0.21 to 0.30]

12. Secondary Outcome: Anti-polyribosylribitol Phosphate (Anti-PRP) and Anti-polysaccharide C (Anti-PSC) Concentration
Description: as for outcome 11
Time Frame: One month after the third dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per milliliter (µg/mL)
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 140 | 142
micrograms per milliliter (µg/mL)
  Anti-PRP (n= 140, 142) | 10.437 [8.398 to 12.970] | 10.473 [8.547 to 12.833]
  Anti-PSC (n= 140, 141) | 6.34 [5.57 to 7.22] | 7.46 [6.67 to 8.34]

13. Secondary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Concentration
Description: Anti-HBs concentrations are given as geometric mean concentrations (GMCs) expressed in milli-international units per milliliter (mIU/mL).
Time Frame: Before vaccination (at Day 0)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 112 | 118
mIU/mL | 24.79 [19.82 to 31.00] | 16.67 [13.52 to 20.56]

14. Secondary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Concentration
Description: as for outcome 13
Time Frame: One month after the third dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 129 | 129
mIU/mL | 372.30 [299.98 to 462.04] | 586.58 [473.80 to 726.21]

15. Secondary Outcome: Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titer
Description: rSBA-MenC titers are given as geometric mean titers (GMTs).
Time Frame: Before vaccination (at Day 0)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 141 | 137
Titer | 4.9 [4.5 to 5.5] | 5.9 [4.9 to 6.9]

16. Secondary Outcome: Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titer
Description: rSBA-MenC titers are given as geometric mean titers (GMTs).
Time Frame: One month after the third dose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 143 | 140
Titer | 1055.9 [859.1 to 1297.7] | 1346.2 [1130.4 to 1603.1]

17. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling and are presented across doses.
Time Frame: During the 4-day follow-up period after any primary vaccination dose
Population: Analysis was performed on the Primary Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 163 | 150
subjects
  Pain | 106 | 100
  Redness | 94 | 123
  Swelling | 91 | 113

18. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Solicited general symptoms assessed include drowsiness, fever, irritability/fussiness and loss of appetite and are presented across doses.
Time Frame: During the 4-day follow-up period after any primary vaccination dose
Population: Analysis was performed on the Primary Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 163 | 150
subjects
  Drowsiness | 111 | 102
  Fever | 89 | 85
  Irritability/fussiness | 128 | 105
  Loss of appetite | 99 | 100

19. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 31 days after each primary vaccination
Population: Analysis was performed on the Primary Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 163 | 150
subjects | 56 | 72

20. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the entire primary vaccination phase
Population: Analysis was performed on the Primary Total Vaccinated Cohort.
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 163 | 150
subjects | 11 | 8

21. Secondary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentration Greater Than or Equal to 0.15 Migrogram Per Milliliter (µg/mL)
Description: Anti-PRP antibody cut-off value assessed was 0.15 migrogram per milliliter (µg/mL).
Time Frame: Prior to (Month 14) and one month after the booster vaccination (Month 15)
Population: Analysis was performed on the Booster ATP cohort for immunogenicity, which included subjects having received 3 vaccine doses during the primary vaccination course and the booster vaccine dose and for whom assay results were available for antibodies against at least one study vaccine antigen component after booster dose administration.
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 133 | 134
subjects
  Pre-booster (n= 133; 130) | 116 | 117
  Post-booster (n= 132; 134) | 132 | 134

22. Secondary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentration Greater Than or Equal to 1.0 Migrogram Per Milliliter (µg/mL)
Description: Anti-PRP antibody cut-off value assessed was 1.0 migrogram per milliliter (µg/mL).
Time Frame: Prior to (Month 14) and one month after the booster vaccination (Month 15)
Population: as for outcome 21
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 133 | 134
subjects
  Pre-booster (n= 133; 130) | 53 | 53
  Post-booster (n= 132; 134) | 132 | 134

23. Secondary Outcome: Number of Subjects With Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titer Greater Than or Equal to the Cut-off Values
Description: rSBA-MenC titer cut-off values assessed include 1:8, 1:32 and 1:128.
Time Frame: Prior to (Month 14) and one month after the booster vaccination (Month 15)
Population: as for outcome 21
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 134 | 137
subjects
  ≥ 1:8 pre-booster (n= 134; 134) | 102 | 117
  ≥ 1:8 post-booster (n= 133; 137) | 132 | 136
  ≥ 1:32 pre-booster (n= 134; 134) | 95 | 115
  ≥ 1:32 post-booster (n= 133; 137) | 132 | 136
  ≥ 1:128 pre-booster (n= 134; 134) | 69 | 85
  ≥ 1:128 post-booster (n= 133; 137) | 131 | 136

24. Secondary Outcome: Number of Subjects With Anti-polysaccharide C (Anti-PSC) Antibody Concentration Greater Than or Equal to the Cut-off Values
Description: Anti-PSC antibody cut-off values assessed include 0.3 micrograms per milliliter (µg/mL) and 2.0 µg/mL.
Time Frame: Prior to (Month 14) and one month after the booster vaccination (Month 15)
Population: as for outcome 21
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 130 | 129
subjects
  ≥ 0.3 µg/mL pre-booster (n= 130; 127) | 74 | 92
  ≥ 0.3 µg/mL post-booster (n= 117; 129) | 116 | 129
  ≥ 2.0 µg/mL pre-booster (n= 130; 127) | 11 | 11
  ≥ 2.0 µg/mL post-booster (n= 117; 129) | 105 | 124

25. Secondary Outcome: Number of Subjects With Anti-hepatitis B Surface Antigen (Anti-HBs) Antibody Concentration Greater Than or Equal to the Cut-off Values
Description: Anti-HBs antibody cut-off values assessed include 10 milli-international units per milliliter (mIU/mL) and 100 mIU/mL.
  Note: the protocol planned an analysis on HBs after the booster dose, but this analysis was not performed as the vaccines administered as booster doses did not contain HBs component.
Time Frame: Prior to (Month 14) the booster vaccination
Population: as for outcome 21
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 125 | 116
subjects
  ≥ 10 mIU/mL pre-booster | 121 | 113
  ≥ 100 mIU/mL pre-booster | 61 | 71

26. Secondary Outcome: Anti-polyribosylribitol Phosphate (Anti-PRP) and Anti-polysaccharide C (Anti-PSC) Concentration
Description: Anti-PRP and anti-PSC concentrations are given as geometric mean concentrations (GMCs) in micrograms per milliliter (µg/mL).
Time Frame: Prior to (Month 14) and one month after the booster vaccination (Month 15)
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per milliliter (µg/mL)
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 133 | 134
micrograms per milliliter (µg/mL)
  anti-PRP pre-booster (n= 133; 130) | 0.706 [0.565 to 0.881] | 0.777 [0.622 to 0.972]
  anti-PRP post-booster (n= 132; 134) | 50.343 [41.627 to 60.884] | 54.625 [45.325 to 65.834]
  anti-PSC pre-booster (n= 130; 127) | 0.42 [0.35 to 0.51] | 0.56 [0.47 to 0.67]
  anti-PSC post-booster (n= 117; 129) | 10.06 [8.14 to 12.45] | 11.31 [9.60 to 13.31]

27. Secondary Outcome: Anti-hepatitis B Surface Antigen (Anti-HBs) Concentration
Description: Anti-HBs concentrations are given as geometric mean concentrations (GMCs) in milli-international units per milliliter (mIU/mL).
  Note: Planned analysis in the protocol of HBs after the booster dose was not performed as booster vaccines did not contain HBs component.
Time Frame: Prior to (Month 14) the booster vaccination
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 125 | 116
mIU/mL | 95.9 [75.6 to 121.5] | 145.6 [112.1 to 189.1]

28. Secondary Outcome: Meningococcal Serogroup C Serum Bactericidal Assay Using Rabbit Complement (rSBA-MenC) Titer
Description: rSBA-MenC titers are given as geometric mean titers (GMTs).
Time Frame: Prior to (Month 14) and one month after the booster vaccination (Month 15)
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 134 | 137
titer
  Pre-booster (n= 134; 134) | 79.3 [56.3 to 111.8] | 147.8 [110.9 to 197.1]
  Post-booster (n= 133; 137) | 4883.1 [3783.1 to 6302.9] | 5288.8 [4244.9 to 6589.4]

29. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms (Local and General)
Description: Solicited local symptoms assessed include pain, redness and swelling. Solicited general symptoms assessed include drowsiness, fever, irritability/fussiness and loss of appetite.
Time Frame: During the 4-day follow-up period following booster vaccination
Population: Analysis was performed on the Booster Total Vaccinated cohort which included all vaccinated subjects for whom data for the booster phase were available.
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 154 | 144
subjects
  Pain | 82 | 98
  Redness | 77 | 109
  Swelling | 67 | 94
  Drowsiness | 33 | 46
  Fever | 43 | 53
  Irritability | 70 | 69
  Loss of appetite | 34 | 50

30. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: as for outcome 19
Time Frame: Within 31 days after the booster vaccination (month 15)
Population: as for outcome 29
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 154 | 144
subjects | 34 | 42

31. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
  Period 1 is defined as 31 days after last primary vaccination until administration of booster dose (Month 14).
  Period 2 is defined as the administration of the booster dose until the end of the study (Month 15).
Time Frame: 31 days after last primary vaccination until administration of booster dose (Month 14) and from the administration of the booster dose until the end of the study (Month 15)
Population: as for outcome 29
Measure: Number; unit: subjects
Arm/Group | Preterm Group | Full-term Group
Number analyzed (Participants) | 154 | 144
subjects
  Period 1 | 10 | 2
  Period 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: For SAEs: the whole study period (Day 0 - Month 15); For frequent adverse events: solicited adverse events a 4-day period after vaccination, unsolicited adverse events a 31-day period after vaccination.
Description: Solicited adverse events after primary and booster vaccination are put as separate adverse events. In the description field of these adverse events it is specified to which vaccination phase they belong.
Arm/Group | Preterm Group | Full-term Group
Serious Adverse Events (participants affected / at risk) | 22/163 | 10/150
Other Adverse Events (participants affected / at risk) | 153/163 | 144/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preterm Group (N=163) | Full-term Group (N=150)
Bronchiolitis (Infections and infestations) | 6 | 2
Pneumonia (Infections and infestations) | 4 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Candidiasis (Infections and infestations) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Meningococcal sepsis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Preterm Group (N=163) | Full-term Group (N=150)
Injection site nodule (General disorders) | 3 | 24
Upper respiratory tract infection (Infections and infestations) | 7 | 11
Vomiting (Gastrointestinal disorders) | 9 | 6
Injection site haematoma (General disorders) | 1 | 9
Pain (General disorders) | 106 | 100 — Within 4 days after primary vaccination
Redness (General disorders) | 94 | 123 — Within 4 days after primary vaccination
Swelling (General disorders) | 91 | 113 — Within 4 days after primary vaccination
Drowsiness (General disorders) | 111 | 102 — Within 4 days after primary vaccination
Fever (General disorders) | 89 | 85 — Within 4 days after primary vaccination
Irritability/fussiness (General disorders) | 128 | 105 — Within 4 days after primary vaccination
Loss of appetite (General disorders) | 99 | 100 — Within 4 days after primary vaccination
Pain (General disorders) | 82/154 | 98/144 — Within 4 days after booster dose
Redness (General disorders) | 77/154 | 109/144 — Within 4 days after booster dose
Swelling (General disorders) | 67/154 | 94/144 — Within 4-days after booster vaccination
Drowsiness (General disorders) | 33/154 | 46/144 — Within 4 days after booster vaccination
Fever (General disorders) | 43/154 | 53/144 — Within 4 days after booster vaccination
Irritability/fussiness (General disorders) | 70/154 | 69/144 — Within 4 days after booster vaccination
Loss of appetite (General disorders) | 34/154 | 50/144 — Within 4 days after booster vaccination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.